CLINICAL TRIAL: NCT03363139
Title: "T790M Mutation Testing in Blood by Different Methodologies"_RING Project
Brief Title: T790M Mutation Testing in Blood by Different Methodologies
Status: Completed | Type: Observational
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 17/03_RING
Record Dates: First submitted 2017-11-24; First posted 2017-12-06 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples in a EDTA tube will be drawn to extract DNA and analyse T790M mutation in NSCLC patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with T790M mutation: Patient who has progressed to Tyrosin Kinase inhibitors and has the mutation of the gen T790M
  Interventions: Drug: Tirosin Kinase Inhibitors

INTERVENTIONS:
Drug: Tirosin Kinase Inhibitors — Patients that received Tyrosin Kinase inhibitors and progressed
  Other Names: TKI

SUMMARY:
Three laboratories will participate in the study. Each laboratory will analyze the same samples by different methodologies according to the flow indicated in figure 1. This design will allow comparing the agreement performance of different methods available for T790M identification in circulating-free DNA isolated from peripheral blood.

DETAILED DESCRIPTION:
Three blood samples per patient will be collected once at the time of progression, assessed by CT Scans according to RECIST criteria v.1.1 and before the patients start a new treatment The blood samples (5-10 mL each) will be collected in one Cell-Free DNA BCT Streck® and 2 PTT EDTA K2 (BECTON DICKINSON) collection tubes.

All samples will be labeled properly with the patient identification number and date of extraction. These samples will be stored and distributed through the 3 participating laboratories until completion of all the analyses, according to the flowchart in Figure 1. These samples will be registered in the samples collection of the Institute of Health Carlos III Registry. These samples will be kept in each participant laboratory after the completion of the RING study and the patient will be informed of that in the patient information sheet and informed consent.

cfDNA will be extracted using as starting volume 1 ml of plasma with a Maxwell® RSC instrument (Promega), using the Maxwell® RSC cfDNA Plasma Kit (MR), as specified by the manufacturer or with a Qiasymphony instrument (Qiagen company). Additionally, for BEAMing analysis, 3 ml of plasma will be used for cfDNA isolation using the the QIAamp® Circulating Nucleic Acid Kit (Qiagen company), following the manufacturer instructions.

Circulating free DNA from peripheral blood sample is an adequate source for T790M resistance mutation testing. However, comparison across different platforms has been scarcely reported. Discordant results for EGFR biomarker testing could impact patient management.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with EGFR mutant, stage IIIB and IV non small cell lung cancer and who have progressed assessed by CT Scans according to RECIST criteria v.1.1 to first or second generation EGFR tyrosine kinase inhibitors (TKIs) (e.g. gefitinib, erlotinib, afatinib) including patients who received a chemotherapy line before TKI treatment. Samples have to be drawn before the patient starts a new treatment,
* Patients have to sign the informed consent of the study
* Patients aged ≥ 18 years.

Exclusion Criteria:

* Patients progressing to third generation EGFR TKIs (e.g. Osimertinib (TKI))
* No possibility of venipuncture.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EGFR mutant non small cell lung cancer patients.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Assess the agreement between qualitative methodologies | At 12 months from the first inclusion
  To evaluate the agreement performance of different methodologies available in Spain for T790M identification in circulating-free DNA isolated from blood collected at the time of progression on a first or second generation TKI

SECONDARY OUTCOMES:
Cost of the different methodologies | At 12 months from the first inclusion
  To compare the cost of the different methodologies
Specificity and sensitivity of each cfDNA method | At 12 months from the first inclusion
  To estimate the specificity and sensitivity of each cfDNA method.

OTHER OUTCOMES:
Turnaround time of different methodologies | At 12 months from the first inclusion
  To compare turnaround time of the different methodologies
Ease of use of different methodologies | At 12 months from the first inclusion
  To compare the ease of use of the different methodologies

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, PhD, Principal Investigator — Hospital Puerta del Hierro
Locations (30):
- Spain (30):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Complejo Hospitalario Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - H. Son Espases, Palma de Mallorca, Mallorca
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - H. Gen. Universitario de Alicante, Alicante
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Instituto Universitario Dexeus, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario de Ciudad Real, Ciudad Real
  - ICO Girona -H. Dr. Josep Trueta, Girona
  - Hospital Clínico San Cecilio, Granada
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Asistencial Universitario de León, León
  - Hospital Lucus Agustí, Lugo
  - H.U. Puerta de Hierro, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Sanchinarro, Madrid
  - H. Carlos Haya, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital La Fe, Valencia
  - H. Gen. Univ. Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Romero A, Jantus-Lewintre E, Garcia-Pelaez B, Royuela A, Insa A, Cruz P, Collazo A, Perez Altozano J, Vidal OJ, Diz P, Cobo M, Hernandez B, Vazquez Estevez S, Benitez G, Guirado M, Majem M, Bernabe R, Ortega AL, Blasco A, Bosch-Barrera J, Jurado JM, Garcia Gonzalez J, Viteri S, Garcia Giron C, Massuti B, Lopez Martin A, Rodriguez-Festa A, Calabuig-Farinas S, Molina-Vila MA, Provencio M. Comprehensive cross-platform comparison of methods for non-invasive EGFR mutation testing: results of the RING observational trial. Mol Oncol. 2021 Jan;15(1):43-56. doi: 10.1002/1878-0261.12832. Epub 2020 Nov 13. PMID 33107189
- See also: Grupo Español de Cáncer de Pulmón — http://www.gecp.org